CLINICAL TRIAL: NCT02240472
Title: Survival and Axillary Recurrence Following Sentinel Node-positive Breast Cancer Without Completion Axillary Lymph Node Dissection - a Randomized Study of Patients With Macrometastases in the Sentinel Node
Brief Title: Sentinel Node Biopsy in Breast Cancer: Omission of Axillary Clearance After Macrometastases. A Randomized Trial.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Cancer Foundation (Other); Nordic Cancer Union (Other)
Responsible Party: Principal Investigator, Jana de Boniface, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENOMAC
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: sentinel node biopsy, lymph node metastasis, survival
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Axillary clearance (No Intervention): Patients in this arm will be treated by completion axillary clearance after a sentinel node biopsy showing 1-2 nodes with macrometastasis
- No axillary clearance (Experimental): Patients in this arm will not undergo further axillary surgery after a sentinel node biopsy showing 1-2 nodes with macrometastasis
  Interventions: Procedure: Omission of axillary clearance

INTERVENTIONS:
Procedure: Omission of axillary clearance — The intervention is the omission of completion axillary clearance after the detection of sentinel node macrometastasis
  Arms: No axillary clearance

SUMMARY:
Since the introduction of sentinel node biopsy in breast cancer, it has become clear that its use is reliable and reproducible. Today, it is clinical routine to not remove further lymph nodes from the axilla (arm pit) in case the sentinel node (which is the first lymph node/s reached by lymphatic flow from the breast) is free of tumor deposits. It is also routine to leave remaining lymph nodes behind in case the sentinel node contains a minimal cluster of tumor cells, called isolated tumor cells (formerly submicrometastasis). Even in slightly larger tumor deposits, so called micrometastasis (up to 2 mm in size), it has been shown that a completion axillary clearance (removal of further lymph nodes from the arm pit) does not contribute to a better survival. Data from a randomized study indicate that it seems safe to omit axillary clearance even if the sentinel node biopsy shows up to 2 nodes with tumor deposits over 2 mm in size (macrometastasis). These studies have changed clinical practice in many countries, however, it is still debated whether it is safe to omit axillary clearance in the case of sentinel node macrometastasis due to under-recruitment in the aforementioned study. The rationale for omitting extensive axillary surgery is the avoidance of postoperative morbidity such as arm lymphedema, loss of sensation, pain and swelling.

The hypothesis is that refraining from axillary clearance in breast cancer patients with 1-2 sentinel nodes with macrometastasis will not worsen breast cancer-specific survival by more than a maximum of 2.5% after 5 years.

This study is a prospective international randomized trial including 3500 patients.

Breast cancer patients without signs of axillary nodal involvement will be eligible for sentinel node biopsy. Those who are found to have up to two sentinel node containing macrometastasis will be informed about this trial Those wishing to participate will be randomized to either undergo further axillary surgery (clearance) or not. Outcome measures are breast cancer-specific survival, disease-free survival, axillary recurrence rate and overall survival.

DETAILED DESCRIPTION:
Details can be found on www.senomac.se

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive breast cancer (T1-T3)
* N0 on palpation
* Preoperative ultrasound performed
* Pathology report shows macrometastasis in 1-2 sentinel lymph nodes
* Patients undergo breast-conserving therapy or mastectomy
* The patient must have provided oral and written consent
* Age ≥ 18 years

Exclusion Criteria:

* Metastases outside of the ipsilateral axilla
* Prior history of invasive breast cancer
* Pregnancy
* Bilateral breast cancer if one side meets exclusion criteria
* Medical contraindication for radiotherapy or systemic treatment
* Inability to absorb or understand the meaning of the study information; for example, through disability, inadequate language skills or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
breast cancer-specific survival | up to 15 years
  death due to breast cancer in both arms measured at a median follow-up of 5, 10 and 15 years

SECONDARY OUTCOMES:
disease-free survival | 5, 10 and 15 years
  Breast cancer recurrence rate in both arms after a median follow-up of 5, 10 and 15 years
axillary recurrence rate | 5, 10 and 15 years
  The rate of axillary relapse in specific after a median follow-up of 5, 10 and 15 years
overall survival | 5, 10 and 15 years
  The rate of overall deaths after a median follow-up of 5, 10 and 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Jana de Boniface, PhD, Principal Investigator — Karolinska Institutet; Jan Frisell, Professor, Study Chair — Karolinska University Hospital; Leif Bergkvist, Professor, Study Chair — Central Hospital Västerås; Yvette Andersson, PhD, Study Chair — Central Hospital Västerås; Lisa Ryden, Professor, Study Chair — Lund University; Malin Sund, Professor, Study Chair — Umeå University Hospital; Olofsson Roger, PhD, Study Chair — Sahlgrenska University Hospital; Johan Ahlgren, PhD, Study Chair — Region Örebro County; Dan Lundstedt, PhD, Study Chair — Sahlgrenska University Hospital; Peer Christiansen, Professor, Principal Investigator — Aarhus University Hospital, Denmark; Tove Tvedskov Filtenborg, MD, Study Chair — Rigshospitalet Copenhagen, Dnmark; Michalis Kontos, PhD, Study Chair — University of Athens; Birgitte Offersen, Professor, Study Chair — University of Aarhus; Thorsten Kühn, Professor, Principal Investigator — Klinikum Esslingen; Toralf Reimer, Professor, Principal Investigator — Universität Rostock; Oreste Gentilini, Principal Investigator — San Raffaele Hospital, Milano; Roland Reitsamer, Principal Investigator — Universitätsklinikum Salzburg
Locations (33):
- Denmark (9):
  - Sygehus Sonderjylland, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Sydvestjysk Sygehus, Esbjerg
  - Sygehus Lillebaelt, Lillebaelt
  - Odense University Hospital, Odense
  - Randers Regionshospitalet, Randers
  - Regionshospitalet Viborg, Viborg
- Athens University Hospital, Athens, Greece
- Sweden (23):
  - Gävle sjukhus, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Hallands sjukhus, Halmstad
  - Helsingborg lasarett, Helsingborg
  - Länssjukhuset Ryhov, Jönköping
  - Kalmar sjukhus, Kalmar
  - Blekinge sjukhuset, Karlskrona
  - Karlstad sjukhus, Karlstad
  - Central Hospital Kristianstad, Kristianstad
  - Linköping University Hospital, Linköping
  - Malmö/Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Skaraborgs sjukhus, Skövde/Lidköping
  - Karolinska University Hospital, Stockholm
  - Southern Gerenal Hospital, Stockholm
  - St. Görans Hospital, Stockholm
  - Sundsvall länssjukhus, Sundsvall
  - Uddevalla sjukhus, Uddevalla
  - Umeå University Hospital, Umeå
  - Akademiska Sjukhuset, Uppsala
  - Varbergs sjukhus, Varberg
  - Västerås Central Hospital, Västerås
  - Västervik Hospital, Västervik

REFERENCES:
- [Derived] Skarping I, Bendahl PO, Szulkin R, Alkner S, Andersson Y, Bergkvist L, Christiansen P, Filtenborg Tvedskov T, Frisell J, Gentilini OD, Kontos M, Kuhn T, Lundstedt D, Vrou Offersen B, Olofsson Bagge R, Reimer T, Sund M, Ryden L, de Boniface J. Prediction of High Nodal Burden in Patients With Sentinel Node-Positive Luminal ERBB2-Negative Breast Cancer. JAMA Surg. 2024 Dec 1;159(12):1393-1403. doi: 10.1001/jamasurg.2024.3944. PMID 39320882
- [Derived] de Boniface J, Appelgren M, Szulkin R, Alkner S, Andersson Y, Bergkvist L, Frisell J, Gentilini OD, Kontos M, Kuhn T, Lundstedt D, Offersen BV, Olofsson Bagge R, Reimer T, Sund M, Christiansen P, Ryden L, Filtenborg Tvedskov T; SENOMAC Trialists' Group. Completion axillary lymph node dissection for the identification of pN2-3 status as an indication for adjuvant CDK4/6 inhibitor treatment: a post-hoc analysis of the randomised, phase 3 SENOMAC trial. Lancet Oncol. 2024 Sep;25(9):1222-1230. doi: 10.1016/S1470-2045(24)00350-4. Epub 2024 Aug 6. PMID 39121881
- [Derived] de Boniface J, Filtenborg Tvedskov T, Ryden L, Szulkin R, Reimer T, Kuhn T, Kontos M, Gentilini OD, Olofsson Bagge R, Sund M, Lundstedt D, Appelgren M, Ahlgren J, Norenstedt S, Celebioglu F, Sackey H, Scheel Andersen I, Hoyer U, Nyman PF, Vikhe Patil E, Wieslander E, Dahl Nissen H, Alkner S, Andersson Y, Offersen BV, Bergkvist L, Frisell J, Christiansen P; SENOMAC Trialists' Group; SENOMAC Trialists' Group. Omitting Axillary Dissection in Breast Cancer with Sentinel-Node Metastases. N Engl J Med. 2024 Apr 4;390(13):1163-1175. doi: 10.1056/NEJMoa2313487. PMID 38598571
- [Derived] Appelgren M, Sackey H, Wengstrom Y, Johansson K, Ahlgren J, Andersson Y, Bergkvist L, Frisell J, Lundstedt D, Ryden L, Sund M, Alkner S, Vrou Offersen B, Filtenborg Tvedskov T, Christiansen P, de Boniface J; SENOMAC Trialists' Group. Patient-reported outcomes one year after positive sentinel lymph node biopsy with or without axillary lymph node dissection in the randomized SENOMAC trial. Breast. 2022 Jun;63:16-23. doi: 10.1016/j.breast.2022.02.013. Epub 2022 Mar 1. PMID 35279508
- [Derived] de Boniface J, Ahlgren J, Andersson Y, Bergkvist L, Frisell J, Lundstedt D, Olofsson Bagge R, Ryden L, Sund M; SENOMAC Trialists' Group. The generalisability of randomised clinical trials: an interim external validity analysis of the ongoing SENOMAC trial in sentinel lymph node-positive breast cancer. Breast Cancer Res Treat. 2020 Feb;180(1):167-176. doi: 10.1007/s10549-020-05537-1. Epub 2020 Jan 27. PMID 31989379
- [Derived] de Boniface J, Frisell J, Andersson Y, Bergkvist L, Ahlgren J, Ryden L, Olofsson Bagge R, Sund M, Johansson H, Lundstedt D; SENOMAC Trialists' Group. Survival and axillary recurrence following sentinel node-positive breast cancer without completion axillary lymph node dissection: the randomized controlled SENOMAC trial. BMC Cancer. 2017 May 26;17(1):379. doi: 10.1186/s12885-017-3361-y. PMID 28549453
- See also: study homepage — http://senomac.se
- Available data/document: Study Protocol — http://senomac.se/Home/study%20protocol.html — Study protocol and patient information (English)

DOCUMENTS (2):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT02240472/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02240472/SAP_001.pdf